CLINICAL TRIAL: NCT00575250
Title: Osteoporosis Education Clinic Study
Brief Title: Education for Osteoporosis in Persons With Existing Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Adelaide (Other)
Collaborators: Osteoporosis SA (Unknown)
Responsible Party: Ms Laura Laslett, University of Adelaide
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2.180405
Record Dates: First submitted 2007-12-17; First posted 2007-12-18 (Estimated); Last update posted 2007-12-18 (Estimated); Status verified 2007-12

CONDITIONS: Osteoporosis
Keywords: Osteoporosis/prevention & control; Osteoporosis Prevention and Self-Management Course; Patient Education/*trends//Questionnaires; Adult//Aged//Middle Aged; Life Style//
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Osteoporosis Prevention and Self-Management Course (4 x 2 1/2 hours)
  Interventions: Behavioral: Osteoporosis Prevention and Self-Management Course
- 2 (Active Comparator): One "introductory" osteoporosis education session (1 x 2 1/2 hours)
  Interventions: Behavioral: Introductory education session on osteoporosis

INTERVENTIONS:
Behavioral: Osteoporosis Prevention and Self-Management Course — Four weekly education sessions of 2 1/2 hours duration, in a group session facilitated by a community nurse and trained lay leader.
  Arms: 1
Behavioral: Introductory education session on osteoporosis — Introductory education session, 1 x 2 1/2 hours in a group session facilitated by a community nurse and trained lay person.
  Arms: 2

SUMMARY:
We wish to investigate whether a weekly, 2½ hour group-based osteoporosis education intervention (the Osteoporosis Prevention and Self-Management Course), is different to one session course (1x 2½ hours) on osteoporosis knowledge, confidence to eat calcium-containing foods, confidence to exercise, and amount of exercise undertaken after three and nine months of follow-up in people aged over 50 years who have already had a bone fracture.

DETAILED DESCRIPTION:
Instruments used to determine change after 3 and 9 months:

Osteoporosis knowledge: Osteoporosis Knowledge Assessment Test (Winzenberg et al. BMC Musculoskelet Disord 2003) Calcium intake: Food frequency questionnaire (Angus et al. J Am Diet Assoc 1989) Calcium and exercise self-efficacy: Osteoporosis Self-Efficacy Scale (Horan et al Res Nurs Health 1998) Physical activity: CHAMPS II (Stewart et al. J Gerontol A Biol Sci Med Sci 2001)

ELIGIBILITY:
Inclusion Criteria:

* Presented to Modbury Hospital's Accident and Emergency Department with a new bone fracture

Exclusion Criteria:

* Residence in nursing home
* Fracture sustained in motor bike, push bike or motor vehicle accident
* Fracture sustained due to high trauma, such as fall from roof or ladder
* Dementia
* Inability to participate in group settings
* Inability to understand spoken English
* Inability to provide informed consent
* Pathological fracture
* Usual place of residence outside South Australia

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2004-01; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Difference between groups at three months on osteoporosis knowledge, confidence in ability to consume calcium and to exercise, actual calcium consumption and exercise levels | Three and nine months

SECONDARY OUTCOMES:
Changes between baseline and three months within each group on osteoporosis knowledge, confidence in the ability to each calcium-containing foods and exercise, and the amount of calcium consumed in foods and exercise undertaken | Three and nine months

CONTACTS AND LOCATIONS:
Overall Officials: Laura L Laslett, MMedSci, Principal Investigator — University of Adelaide; Julian D McNeil, PhD FRACP, Study Chair — University of Adelaide
Locations (1):
- Modbury Hospital, Modbury, Adelaide, South Australia, Australia